CLINICAL TRIAL: NCT04488237
Title: Effect of Vitamin D Administration on Methotrexate Adverse Effects in Patients With Acute Lymphoblastic Leukemia
Brief Title: Vitamin D and Methotrexate Adverse Effects
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Magy Ibrahim Anis Rizkallah, Demonstrator of cancer biology, Assiut University
Other Study IDs: MTX side effects and VitD
Record Dates: First submitted 2020-07-23; First posted 2020-07-27 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: methotrexate; vitamin D
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Vitamin D

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Vitamin D — oral administration of Vitamin D in patients with acute leukemia treated with methotrexate

SUMMARY:
Since methotrexate toxicity represents a major problem in patients treating with cancer and there are few studies about the role of vitamin D in the pathogenesis of this toxicity, so the aim of the present study is investigation of the effect of vitamin D administration on methotrexate toxicity such as oral ulcerations, bone marrow toxicity as well as renal and hepatic toxicity also the role of inflammatory mediators and oxidative stress markers in methotrexate toxicity will be evaluated, taking in consideration the dose of leucovorin rescue.

DETAILED DESCRIPTION:
Leukemia is a type of blood cancer that affects the body's white blood cells (WBCs). White blood cells help fight infection and protect the body against disease, but in leukemia, some of the white blood cells turn cancerous and don't work as they should. As more cancerous cells form in the blood and bone marrow (spongy tissue inside the bones), there's less room for healthy cells .

The different types of leukemia can be either acute (fast growing) or chronic (slow growing). Acute lymphoblastic leukemia (ALL) happens when the body makes too many lymphoblasts (a type of white blood cell). It's the most common type of childhood cancer.

Treatment outcome of acute leukemia has been improved recently using Methotrexate . Side effects of methotrexate usually in the form of ulcerative stomatitis, leukopenia (lower amount of white blood cells), nausea, abdominal discomfort, and elevated liver and kidney function tests. Identifying risk factors leading to these side effects would be valuable to develop preventive interventions and improve quality of life for these young patients.

Studies revealed a relationship between vitamin D deficiency and adverse reactions of chemotherapy in cancer patients. This vitamin is important in many physiological processes in the body as bone mineralization and immune regulations . A human body produces vitamin D as a response to sun exposure. A person can also boost their vitamin D intake through certain foods or supplements. .

Previous literature showed that receptors for vitamin D expressed in the mucosa and so there is a relationship between vitamin D deficiency and increase inflammation and impairment of mucosa .

Vitamin D is a fat-soluble vitamin that not only regulates calcium absorption and bone metabolism, but can also regulate cell proliferation, differentiation and the immune response, vitamin D insufficiency/deficiency is associated with poor clinical outcome and significantly worse progression free survival of patients from leukemia and lymphoma.

Calcium is the most abundant element in the human body and is essential for life. It has a key role in many physiological processes including skeletal mineralization, muscle contraction, nerve impulse transmission, blood clotting, and hormone secretion . 1, 25-Dihydroxyvitamin D3 the active form of vitamin D plays major role in intestinal calcium absorption, Calcium homeostasis is also regulated by parathyroid hormone.

Patients with acute lymphoblastic leukemia may be at risk of vitamin D deficiency because of impaired vitamin intake and sunlight exposure .

ELIGIBILITY:
Inclusion Criteria:

1. Patients with acute lymphoblastic leukemia who do not start treatment course with methotrexate.
2. Both sex will be included.
3. Age group (1 -12 years)

Exclusion Criteria:

1. Patients with other type of cancer beside ALL.
2. Patients with renal, hepatic or hematological diseases.

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: cases include patients with acute leumphoblastic leukemia recieving methotrexate in treatment protocol
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Effect of vitamin D administration on methotrexate adverse effects in patients with acute lymphoblastic leukemia | 1 to 2 years according to the availability of the cases
  Since methotrexate toxicity represents a major problem in patients treating with cancer and there are few studies about the role of vitamin D in the pathogenesis of this toxicity, so the aim of the present study is investigation of the effect of vitamin D administration on methotrexate toxicity such as oral ulcerations, bone marrow toxicity as well as renal and hepatic toxicity also the role of inflammatory mediators and oxidative stress markers in methotrexate toxicity will be evaluated, taking in consideration the dose of leucovorin rescue.

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Hamdy Abdel-Raheem, Phd, Study Director — Assiut University; Mohammed Mostafa Elbadr, Phd, Study Director — Assiut University; Nivin Abdel-Azim Abdel-Rehim, Phd, Study Director — Assiut University

REFERENCES:
- [Background] Hunger SP, Lu X, Devidas M, Camitta BM, Gaynon PS, Winick NJ, Reaman GH, Carroll WL. Improved survival for children and adolescents with acute lymphoblastic leukemia between 1990 and 2005: a report from the children's oncology group. J Clin Oncol. 2012 May 10;30(14):1663-9. doi: 10.1200/JCO.2011.37.8018. Epub 2012 Mar 12. PMID 22412151
- [Background] Anand A, Singh S, Sonkar AA, Husain N, Singh KR, Singh S, Kushwaha JK. Expression of vitamin D receptor and vitamin D status in patients with oral neoplasms and effect of vitamin D supplementation on quality of life in advanced cancer treatment. Contemp Oncol (Pozn). 2017;21(2):145-151. doi: 10.5114/wo.2017.68623. Epub 2017 Jun 30. PMID 28947884
- [Background] Oosterom N, Dirks NF, Heil SG, de Jonge R, Tissing WJE, Pieters R, van den Heuvel-Eibrink MM, Heijboer AC, Pluijm SMF. A decrease in vitamin D levels is associated with methotrexate-induced oral mucositis in children with acute lymphoblastic leukemia. Support Care Cancer. 2019 Jan;27(1):183-190. doi: 10.1007/s00520-018-4312-0. Epub 2018 Jun 19. PMID 29922939
- [Background] Lalla RV, Choquette LE, Feinn RS, Zawistowski H, Latortue MC, Kelly ET, Baccaglini L. Multivitamin therapy for recurrent aphthous stomatitis: a randomized, double-masked, placebo-controlled trial. J Am Dent Assoc. 2012 Apr;143(4):370-6. doi: 10.14219/jada.archive.2012.0179. PMID 22467697
- [Background] Crew KD, Shane E, Cremers S, McMahon DJ, Irani D, Hershman DL. High prevalence of vitamin D deficiency despite supplementation in premenopausal women with breast cancer undergoing adjuvant chemotherapy. J Clin Oncol. 2009 May 1;27(13):2151-6. doi: 10.1200/JCO.2008.19.6162. Epub 2009 Apr 6. PMID 19349547
- [Background] Fakih MG, Trump DL, Johnson CS, Tian L, Muindi J, Sunga AY. Chemotherapy is linked to severe vitamin D deficiency in patients with colorectal cancer. Int J Colorectal Dis. 2009 Feb;24(2):219-24. doi: 10.1007/s00384-008-0593-y. Epub 2008 Oct 2. PMID 18830610